CLINICAL TRIAL: NCT02075827
Title: Metabolic Response to Playing Video Games: Two Arm Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UCL0326011
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Appetite and General Nutritional Disorders; Sedentary Lifestyle
Keywords: Appetite, metabolism, sedentary behaviour, stress response
MeSH Terms: conditions — Sedentary Behavior; Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problem-solving video game (Active Comparator): Playing the video game 'Little Big Planet'
  Interventions: Behavioral: Little Big Planet
- Competitive video game (Experimental): Playing the video game 'Call of Duty'
  Interventions: Behavioral: Competitive video game

INTERVENTIONS:
Behavioral: Competitive video game — 1 hour playing video game
  Other Names: 'Call of Duty' (Activision)
  Arms: Competitive video game
Behavioral: Little Big Planet — 1 hour playing video game
  Other Names: Little Big Planet (Sony Computer Entertainment
  Arms: Problem-solving video game

SUMMARY:
Previous studies have shown that subjects who play video games are prone to consume larger quantities of food than subjects who are simply resting. This is believed to be due to the development of a stress response in the video games group, resulting in increased fuel metabolism. However, it was shown that the energy intake of the two groups showed no correlation with the subjects' appetite/hunger, which was identical in both groups.

The investigators propose to explore this issue further by comparing the effects of different types of video games on metabolism, using a randomized controlled trial. In this study, they will compare the stress levels, heart rate, blood pressure, appetite/mood, energy consumption, grip strength, memory and saliva cortisol, leptin and ghrelin levels of subjects playing (a) competitive and (b) problem-solving video games. Measurements will be taken preceding, during and after the 1 hour intervention. Following the intervention, participants will be offered savoury and sweet foods/drinks, which will allow us to assess their appetite preferences and caloric intake.

The investigators first aim is to determine whether there is a significant difference in stress levels, eating habits and energy metabolism in the two groups. Our second aim is to determine whether there is a difference in glucose distribution to the muscles and brain between the two groups.

DETAILED DESCRIPTION:
The investigators study is designed to test experimentally whether different kinds of video game generate different types of metabolic response. The exposure comprises one-hour of video game playing, with 36 young men randomized to each group (ie 72 in total).

Prior to the exposure, they will collect baseline data on heart rate, blood pressure, anthropometry (weight, height, waist girth), grip strength and cognitive function (memory test), as well as appetite/mood by visual analogue scale (VAS). The investigators will also collect a baseline saliva sample to assess hormones associated with stress (cortisol) or satiety (leptin, ghrelin). The subject will arrive after and overnight fast and will be given a standardised breakfast. After these baseline data are collected, the randomization envelope will be opened and the subject assigned to his group.

Heart rate will be monitored continuously during the study. At 20 and 40 minutes during the intervention, as well as when it ceases at 60 minutes, the investigators will collect further data on blood pressure and appetite/mood by VAS. At 60 minutes, the investigators will repeat measurement of memory and grip strength, and collect a second saliva sample.

For 20 minutes after the end of the intervention, the subject will be allowed to rest, reading magazines, and will be able to select from a range of snack foods (savoury, sweet, fruit), and drinks (sweetened beverages, water). Consumption of calories will be calculated. At the end of this period, final measurements of blood pressure and VAS will be collected, and the subject will depart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males with BMI <25 kg/m2

Exclusion Criteria:

* smoking
* a significant weight change (>3kg) within the previous three months
* any psychiatric disorder
* uncontrolled hypertension
* coronary heart disease
* heart failure
* central/peripheral arteriopathies
* excessive alcohol consumption (<21 units/week).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Food intake | At end of 1-hour video game intervention
  Subjects will be offered a selection of snacks and drinks over a 20 minute period, and their rates of food intake will be calculated

SECONDARY OUTCOMES:
Blood pressure | At 20, 40 and 60 minutes of intervention, and after 20 minutes rest post-intervention
  Blood pressure will be measured in duplicate at 1 minute intervals by digital instrument
Heart rate | Continuously, starting during baseline period, from 0 to 60 minutes during intervention, and for 20 minutes post-intervention rest period
  Heart rate will be measured using a polar digital heart rate monitor
Salivary leptin | After 60 minutes from start of intervention
  Salivary leptin will be analysed using ELISA
Salivary ghrelin | After 60 minutes from start of intervention
  Salivary ghrelin will be assessed using ELISA
Salivary cortisol | After 60 minutes from start of intervention
  Salivary cortisol will be assessed using ELISA
Visual analogue scale | At 20, 40 and 60 minutes of intervention, and after 20 minutes rest post-intervention
  Visual analogue scale will be used to collect subjective data on mood and appetite
Grip strength | After 60 minutes from start of intervention
  Grip strength will be assessed by hand-grip dynamometer, using the average of three measurements for each arm
Memory recall | After 60 minutes from start of intervention
  Subjects will be shown images for a set time to allow memorization, and then be given another set time to recall as many of these images as possible

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan CK Wells, PhD, Principal Investigator — UCL Institute of Child Health
Locations (1):
- UCL Institute of Child Health, London, United Kingdom

REFERENCES:
- [Background] Siervo M, Sabatini S, Fewtrell MS, Wells JC. Acute effects of violent video-game playing on blood pressure and appetite perception in normal-weight young men: a randomized controlled trial. Eur J Clin Nutr. 2013 Dec;67(12):1322-4. doi: 10.1038/ejcn.2013.180. Epub 2013 Oct 2. PMID 24084510